CLINICAL TRIAL: NCT02695810
Title: Effect of Dapagliflozin, Metformin and Physical Activity on Glucose Variability, Body Composition and Cardiovascular Risk in Pre-diabetes
Brief Title: The PRE-D Trial: Effect of Dapagliflozin, Metformin and Physical Activity in Pre-diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: The Novo Nordic Foundation (Other); Rigshospitalet, Denmark (Other); AstraZeneca (Industry); Bayer (Industry)
Responsible Party: Principal Investigator, Kristine Færch, Senior Researcher, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-001552-30
Record Dates: First submitted 2016-02-09; First posted 2016-03-01 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Prediabetic State; Obesity
MeSH Terms: conditions — Prediabetic State; Obesity | interventions — dapagliflozin; Metformin; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dapagliflozin (Experimental): Dapagliflozin, 10 mg per day
  Interventions: Drug: Dapagliflozin
- Metformin (Active Comparator): Metformin, 2 x 850 mg per day
  Interventions: Drug: Metformin
- Exercise (Active Comparator): Exercise, interval training
  Interventions: Behavioral: Exercise
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg per day as monotherapy for 13 weeks
  Other Names: Forxiga, AstraZeneca
  Arms: Dapagliflozin
Drug: Metformin — 2 x 850 mg per day as monotherapy for 13 weeks
  Other Names: Aurobindo, Orion Pharma
  Arms: Metformin
Behavioral: Exercise — Interval training, 5 times per week, 30 min per session
  Arms: Exercise

SUMMARY:
The overall objective is to compare the short-term (3 months) effectiveness of three glucose-lowering interventions (dapagliflozin, metformin and physical activity) on glucose variability, body composition, and cardiometabolic risk factors in overweight or obese individuals with pre-diabetes (HbA1c 5.7-6.4% / 39-47 mmol/mol).

DETAILED DESCRIPTION:
Different medical therapies and lifestyle modification for the prevention of type 2 diabetes have yet to be compared head-to-head in individuals with pre-diabetes. This research project will compare different glucose-lowering interventions in overweight and obese individuals with HbA1c levels in the pre-diabetic range.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c: from ≥5.7% (39 mmol/mol) to ≤6.4% (47 mmol/mol)
* Age: from ≥30 to ≤70 years of age
* BMI ≥25 kg/m2

Exclusion Criteria:

* Uncontrolled medical issues including but not limited to cardiovascular pulmonary, rheumatologic, hematologic, oncologic, infectious, gastrointestinal or psychiatric disease; diabetes or other endocrine disease; immunosuppression;
* Current treatment with hormones which affect glucose metabolism;
* Current treatment with loop diuretics or thiazolidinediones;
* Current treatment with beta blockers or peroral steroids;
* Bariatric surgery within the past 2 years;
* Impaired renal function defined as an estimated GFR<60 ml/min/1.73m2;
* Neurogenic bladder disorders;
* Alcohol/drug abuse or in treatment with disulfiram (Antabus) at time of inclusion;
* Pregnant or lactating women;
* Fertile women not using birth control agents including oral contraceptives, gestagen injection, subdermal implants, hormonal vaginal ring, transdermal application, or intra-uterine devices;
* Allergic to one or more of the medications used in the study;
* Concomitant participation in other intervention study;
* Unable to understand the informed consent and the study procedures.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2019-01-13 (Actual)

PRIMARY OUTCOMES:
Mean amplitude of glycaemic excursions (MAGE) as assessed by continuous glucose monitoring | Change from baseline to 13 weeks and 26 weeks

SECONDARY OUTCOMES:
Intra-day glycaemic variability as assessed by continuous overall net glycaemic action (CONGA) | Change from baseline to 13 weeks and 26 weeks
Daily time spent above different glucose concentrations ( e.g. >6.1 mmol/L, >7.0 mmol/L, >7.8 mmol/L, and >11.1 mmol/L) | Change from baseline to 13 weeks and 26 weeks
HbA1c | Change from baseline to 13 weeks and 26 weeks
Glucose concentrations during OGTT | Change from baseline to 13 weeks and 26 weeks
Insulin secretion as assessed by the insulinogenic index | Change from baseline to 13 weeks and 26 weeks
Insulin sensitivity as assessed by the insulin sensitivity index | Change from baseline to 13 weeks and 26 weeks
Body weight (kg) | Change from baseline to 13 weeks and 26 weeks
Body fat (%) as assessed by DEXA scan | Change from baseline to 13 weeks and 26 weeks
Cardiorespiratory fitness as assessed by maximal oxygen uptake (VO2 max) | Change from baseline to 13 weeks and 26 weeks
Respiratory exchange ratio (RER) as assessed by indirect calorimetry | Change from baseline to 13 weeks and 26 weeks
Basal metabolic rate (BMR) as assessed by indirect calorimetry | Change from baseline to 13 weeks and 26 weeks
Time spent sedentary and in moderate-to-vigorous physical activity intensity as assessed by accelerometer | Change from baseline to 13 weeks and 26 weeks
Systolic and diastolic blood pressure | Change from baseline to 13 weeks and 26 weeks
Plasma lipids | Change from baseline to 13 weeks and 26 weeks
Number of self-reported adverse events and side effects | Change from baseline to 13 weeks and 26 weeks
Self-rated health and quality of life as assessed by questionnaire | Change from baseline to 13 weeks and 26 weeks
Sleep habits as assessed by questionnaire | Change from baseline to 13 weeks and 26 weeks
Dietary intake as assessed by a food diary | Change from baseline to 13 weeks and 26 weeks
Adherence to the different interventions as assessed by number of tablets returned or number of training passes completed | Change from baseline to 13 weeks and 26 weeks
Responsiveness to interventions in individuals with different glucose tolerance status (impaired fasting glycaemia vs. impaired glucose tolerance) | Change from baseline to 13 weeks and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marit E Jørgensen, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center A/S, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perreault L, Faerch K. Approaching pre-diabetes. J Diabetes Complications. 2014 Mar-Apr;28(2):226-33. doi: 10.1016/j.jdiacomp.2013.10.008. Epub 2013 Oct 28. PMID 24342268
- [Background] Faerch K, Hulman A, Solomon TP. Heterogeneity of Pre-diabetes and Type 2 Diabetes: Implications for Prediction, Prevention and Treatment Responsiveness. Curr Diabetes Rev. 2016;12(1):30-41. doi: 10.2174/1573399811666150416122903. PMID 25877695
- [Background] Faerch K, Vistisen D, Johansen NB, Jorgensen ME. Cardiovascular risk stratification and management in pre-diabetes. Curr Diab Rep. 2014 Jun;14(6):493. doi: 10.1007/s11892-014-0493-1. PMID 24743942
- [Derived] Hulman A, Foreman YD, Brouwers MCGJ, Kroon AA, Reesink KD, Dagnelie PC, van der Kallen CJH, Greevenbroek MMJV, Faerch K, Vistisen D, Jorgensen ME, Stehouwer CDA, Witte DR. Towards precision medicine in diabetes? A critical review of glucotypes. PLoS Biol. 2021 Mar 11;19(3):e3000890. doi: 10.1371/journal.pbio.3000890. eCollection 2021 Mar. PMID 33705389
- [Derived] Faerch K, Blond MB, Bruhn L, Amadid H, Vistisen D, Clemmensen KKB, Vaino CTR, Pedersen C, Tvermosegaard M, Dejgaard TF, Karstoft K, Ried-Larsen M, Persson F, Jorgensen ME. The effects of dapagliflozin, metformin or exercise on glycaemic variability in overweight or obese individuals with prediabetes (the PRE-D Trial): a multi-arm, randomised, controlled trial. Diabetologia. 2021 Jan;64(1):42-55. doi: 10.1007/s00125-020-05306-1. Epub 2020 Oct 16. PMID 33064182
- [Derived] Faerch K, Amadid H, Nielsen LB, Ried-Larsen M, Karstoft K, Persson F, Jorgensen ME. Protocol for a randomised controlled trial of the effect of dapagliflozin, metformin and exercise on glycaemic variability, body composition and cardiovascular risk in prediabetes (the PRE-D Trial). BMJ Open. 2017 Jun 6;7(5):e013802. doi: 10.1136/bmjopen-2016-013802. PMID 28592573
- See also: Steno Diabetes Center — http://steno.dk/